CLINICAL TRIAL: NCT03050775
Title: Comparing Patient Temperatures in Adults During Lower Spinal Surgery Using Either a Heated Ventilator Circuit or a Standard Ventilator Circuit With a Heat-Moisture Exchanger
Brief Title: Evaluating Adult Patient Temperatures During Lower Spinal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Westmed, Inc. (Unknown)
Responsible Party: Principal Investigator, Jean M. Guyer, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 15-001604; UL1TR000135 (NIH)
Record Dates: First submitted 2017-02-09; First posted 2017-02-13 (Actual); Results first posted 2018-05-07 (Actual); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Hypothermia
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Intervention Model Description: randomized, trial (treatment or no treatment)
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients were randomly assigned to either the treatment group or the control group prior to surgery. Group randomization was performed using a randomization schedule prepared by the Division of Clinical Statistics with patients randomized in blocks of four. For consented and enrolled patients on the day of surgery in the admit areas, a participant was assigned the next sequential participant ID number and the appropriate sealed envelope was opened to reveal the participant's randomized intervention. This occurred before the patient was transferred to the operating suite. Individuals who performed data analysis were blinded to treatment group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Heated Ventilator Circuit (Experimental): Heated and humidified inspired gases using the ANAPOD™ Heat and Humidification System (Westmed; Tucson, Arizona, USA) circuit prior to induction of general anesthesia in addition to standard ventilation and temperature management.
  Interventions: Device: Heated Ventilator Circuit
- Standard Ventilator Circuit (Active Comparator): Standard ventilation and temperature management.
  Interventions: Device: Standard Ventilator Circuit

INTERVENTIONS:
Device: Heated Ventilator Circuit — active heat and humidification during anesthesia by warming inspire gases without a heat-moisture exchanger
  Other Names: ANAPOD™ Heat and Humidification System
  Arms: Heated Ventilator Circuit
Device: Standard Ventilator Circuit — no active heat and humidification during anesthesia
  Other Names: Thermovent 600; Portex
  Arms: Standard Ventilator Circuit

SUMMARY:
The purpose of this study is to evaluate patients' temperatures after using one of two ventilator circuits (breathing systems): the ANAPOD™ Heat and Humidification System (ANAPOD™ system) or the standard ventilator circuit with a heat-moisture exchanger (standard ventilator). The ANAPOD™ system will provide additional heat and humidity to patients through their breathing tube while the standard ventilator will not. The investigators are doing this research study to find out if the ventilator circuit providing additional heat and humidity will keep patients warmer during surgery and after surgery.

DETAILED DESCRIPTION:
Patients were randomly assigned to either the treatment group or the control group prior to surgery. Prior to induction, patients in the control group were given inspiratory gas at ambient air temperature (20-22 degrees Celsius) and patients in the treatment group were given inspiratory gas at warmed temperatures (40-41 degrees Celsius). All patients were induced with general anesthesia in the supine position and repositioned prone following endotracheal intubation and placement of an esophageal stethoscope with a temperature sensor, as per usual hospital practice. Esophageal temperatures were recorded within 30 minutes of the baseline esophageal temperature and every 10 minutes thereafter for the first hour post-induction. All patients had a blanket and forced air warming applied to their lower extremities and upper back at 43 degrees Celsius after draping. All patients had esophageal temperature measurements recorded every 30 minutes until the patient was repositioned supine. Core temperatures were recorded four hours post-induction for those patients reaching that timeframe.

ELIGIBILITY:
Inclusion Criteria:

* Elective spine surgery anticipated greater than three hours in duration
* Posterior approach
* An operative site between lumbar one and sacral one
* Involving two or more levels with fusion and/or instrumentation and/or revisions
* American Society of Anesthesiologists (ASA) Status of I-III

Exclusion Criteria:

* Patients with a tracheostomy
* Preoperative temperature >38°C or <36°C on the day of surgery
* Active infection or erythema to the back
* White blood cell count greater than 10,500/microliter (mcL)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-08-28 (Actual); Primary Completion 2017-02-05 (Actual); Study Completion 2017-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean M Guyer, DNP, Principal Investigator — Mayo Clinic

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Heated Ventilator Circuit | Standard Ventilator Circuit
Started | 35 | 35
Completed | 35 | 35
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: One subject in the standard group was not included in any of the analyses as this subject's intraoperative temperature was unavailable as part of the anesthetic record.
Groups:
- Total: Total of all reporting groups
Arm/Group | Heated Ventilator Circuit | Standard Ventilator Circuit | Total
Number analyzed (Participants) | 35 | 34 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: One subject in the standard group was not included in any of the analyses as this subject's intraoperative temperature was unavailable as part of the anesthetic record.
  years | 63 (11) | 61 (12) | 62 (11)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One subject in the standard group was not included in any of the analyses as this subject's intraoperative temperature was unavailable as part of the anesthetic record.
  Participants
    Female | 18 | 16 | 34
    Male | 17 | 18 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: One subject in the standard group was not included in any of the analyses as this subject's intraoperative temperature was unavailable as part of the anesthetic record.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 34 | 32 | 66
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants] — Population: One subject in the standard group was not included in any of the analyses as this subject's intraoperative temperature was unavailable as part of the anesthetic record.
  Participants
    United States | 35 | 34 | 69
BMI [Mean (Standard Deviation); unit: kg/m^2] — Population: One subject in the standard group was not included in any of the analyses as this subject's intraoperative temperature was unavailable as part of the anesthetic record.
  kg/m^2 | 28.21 (4.61) | 29.17 (5.90) | 28.69 (5.25)
American Society of Anesthesiologists (ASA) Status [Count of Participants; unit: Participants] — The ASA physical status classification system is a system for assessing the fitness of patients before surgery. There are six categories in the classification system, the higher the number, the more severe illness is indicated. I=normal healthy patient, II=patient with mild systemic disease, III=a patient with severe systemic disease, IV=a patient with severe systemic disease that is a constant threat to life, V=a moribund patient who is not expected to survive without the operation, VI=a declared brain-dead patient whose organs are being removed for donor purposes. Population: One subject in the standard group was not included in any of the analyses as this subject's intraoperative temperature was unavailable as part of the anesthetic record.
  Participants
    ASA I or II | 22 | 21 | 43
    ASA III | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Core Body Temperature
Description: Core body temperature will be taken in the esophagus. The last recorded esophageal temperature will be used for surgeries not reaching 3 hours duration.
Time Frame: Approximately four hours post-induction of general anesthesia (or last recorded temperature)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | Heated Ventilator Circuit | Standard Ventilator Circuit
Number analyzed (Participants) | 35 | 34
degrees Celsius | 36.8 (0.2) | 36.8 (0.2)
Statistical Analysis 1: Comparison: Heated Ventilator Circuit vs Standard Ventilator Circuit; Test type: Superiority; p = 0.807, t-test, 2 sided
Statistical Analysis 2: Comparison: Heated Ventilator Circuit vs Standard Ventilator Circuit; Test type: Superiority; p = 0.358, ANCOVA; Mean Difference (Final Values) = 0.076, 95% CI 2-sided [-0.085 to 0.237]

2. Secondary Outcome: Intraoperative Core Temperatures Post-induction
Description: Core body temperature will be taken in the esophagus after general anesthesia induction.
Time Frame: Approximately 30 minutes, 60 minutes, 120 minutes post-induction of general anesthesia
Population: One subject in the standard group was not included in any of the analyses as this subject's intraoperative temperature was unavailable as part of the anesthetic record.
  Data was obtained from 33 subjects in the treatment group at 60 minutes post-induction.
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | Heated Ventilator Circuit | Standard Ventilator Circuit
Number analyzed (Participants) | 35 | 34
degrees Celsius
  ~30 minutes | 36.1 (0.5) | 36.1 (0.4)
  ~60 minutes: number analyzed (Participants) | 33 | 34
  ~60 minutes | 35.8 (0.6) | 35.8 (0.5)
  ~120 minutes | 36.1 (0.5) | 36.1 (0.4)
Statistical Analysis 1: Comparison: Heated Ventilator Circuit vs Standard Ventilator Circuit; ~30 minutes post-induction; Test type: Superiority; p = 0.823, t-test, 2 sided; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.3 to 0.2]
Statistical Analysis 2: Comparison: Heated Ventilator Circuit vs Standard Ventilator Circuit; ~60 minutes post-induction. Data was obtained from 33 subjects in the treatment group; Test type: Superiority; p = 0.853, t-test, 2 sided; Median Difference (Final Values) = 0.0, 95% CI 2-sided [-0.2 to 0.3]
Statistical Analysis 3: Comparison: Heated Ventilator Circuit vs Standard Ventilator Circuit; ~120 minutes post-induction; Test type: Superiority; p = 0.986, t-test, 2 sided; Median Difference (Final Values) = 0.0, 95% CI 2-sided [-0.2 to 0.2]

3. Secondary Outcome: Number of Subjects With Post-operative Shivering
Description: Shivering in the post-anesthesia care unit will be assessed using the Bedside Shivering Assessment Scale. This is a 4 point scale and rate shivering as the following: absent, mild, moderate, or severe. Only the highest degree of patient shivering was used in the analysis.
Time Frame: Approximately 2 hours after completion of the surgery
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Heated Ventilator Circuit | Standard Ventilator Circuit
Number analyzed (Participants) | 35 | 34
Participants
  Post-operative shivering | 8 | 5
  No post-operative shivering or not assessed | 27 | 29
Statistical Analysis 1: Comparison: Heated Ventilator Circuit vs Standard Ventilator Circuit; Post-operative shivering observed; Test type: Superiority; p = 0.540, Fisher Exact; Odds Ratio (OR) = 1.7, 95% CI 2-sided [0.5 to 5.9]

4. Secondary Outcome: Hospital Length of Stay
Description: Number of days in the hospital
Time Frame: Surgery to hospital discharge
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: number of days
Arm/Group | Heated Ventilator Circuit | Standard Ventilator Circuit
Number analyzed (Participants) | 35 | 34
number of days | 3 [2 to 5] | 3 [2 to 5]
Statistical Analysis 1: Comparison: Heated Ventilator Circuit vs Standard Ventilator Circuit; Test type: Superiority; p = 0.672, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0, 95% CI 2-sided [-1 to 1]

5. Secondary Outcome: Overall Post-operative Temperature
Description: Temperature at Post Anesthesia Care Unit (PACU) arrival.
Time Frame: PACU arrival
Population: One subject in the standard group was not included in any of the analyses as this subject's intraoperative temperature was unavailable as part of the anesthetic record.
  Data was obtained from 32 subjects in the treatment group.
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | Heated Ventilator Circuit | Standard Ventilator Circuit
Number analyzed (Participants) | 32 | 34
degrees Celsius | 36.6 (0.4) | 36.6 (0.4)
Statistical Analysis 1: Comparison: Heated Ventilator Circuit vs Standard Ventilator Circuit; Data was obtained from 32 subjects in the treatment group; Test type: Superiority; p = 0.571, t-test, 2 sided; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.2 to 0.1]

6. Secondary Outcome: Number of Participants With Transfusion Within 48 Hours of Surgery
Description: Requirement of blood transfusion within 48 hours of surgery
Time Frame: Within 48 hours of surgery
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Heated Ventilator Circuit | Standard Ventilator Circuit
Number analyzed (Participants) | 35 | 34
Participants
  No transfusion | 21 | 23
  Transfusion | 14 | 11
Statistical Analysis 1: Comparison: Heated Ventilator Circuit vs Standard Ventilator Circuit; Test type: Superiority; p = 0.619, Fisher Exact; Odds Ratio (OR) = 1.4, 95% CI 2-sided [0.5 to 3.7]

7. Secondary Outcome: Estimated Blood Loss
Description: The estimated blood loss per case was determined by the anesthesia provider by measuring the volume of blood in the suction canister while taking into account the amount of irrigation solution used.
Time Frame: duration of surgery
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: milliters
Arm/Group | Heated Ventilator Circuit | Standard Ventilator Circuit
Number analyzed (Participants) | 35 | 34
milliters | 450 [250 to 1000] | 425 [237.5 to 771.75]
Statistical Analysis 1: Comparison: Heated Ventilator Circuit vs Standard Ventilator Circuit; Test type: Superiority; p = 0.404, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 75, 95% CI 2-sided [-100 to 250]

ADVERSE EVENTS:
Time Frame: 30 days.
Description: One subject in the standard group was not included in any of the analyses as this subject's intraoperative temperature was unavailable as part of the anesthetic record.
Arm/Group | Heated Ventilator Circuit | Standard Ventilator Circuit
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/34
Other Adverse Events (participants affected / at risk) | 5/35 | 3/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Heated Ventilator Circuit (N=35) | Standard Ventilator Circuit (N=34)
Infection (Infections and infestations) | 4 (4) | 3 (3)
Blood clot (Blood and lymphatic system disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was not blinded; investigators were unable to verify exact placement of the esophageal temperature probe; post-op shivering assessments and both OR and ANAPOD temperatures were not consistently recorded at regular intervals.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-26): https://cdn.clinicaltrials.gov/large-docs/75/NCT03050775/Prot_SAP_000.pdf